CLINICAL TRIAL: NCT00918801
Title: Pilot Study of Hippocampal Function in T1DM
Brief Title: Pilot Study of Hippocampal Function in Type 1 Diabetes Mellitus (T1DM)
Acronym: ASSET
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0786
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM; MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes Mellitus: Adolescents ages 13-18 with T1DM
- Non Controls: Healthy adolescents ages 13-18 without T1DM

SUMMARY:
This study is an expansion of a previous study done to determine how thinking skills relate to hypoglycemia (low blood sugar) and certain regions of the brain in children and adolescents. In this study, the investigators are testing thinking skills and measuring brain activity in adolescents with and without type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 18
* Right handed
* Diagnosis of Type 1 Diabetes OR normal sibling control
* If diabetic, then diagnosis for at least 2 years

Exclusion Criteria:

* Pregnant or lactating
* Chronic disease other than well-controlled asthma, or Hashimoto's thyroiditis.
* Other current serious medical illness
* Co-morbid psychiatric illness
* Co-morbid neurological illness
* Pre-maturity at birth
* Contraindication to MRI scan
* orthodontic braces.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young adults will be piloted in a sample of diabetic and non-diabetic adolescents ages 13-18.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2007-04; Primary Completion 2013-12 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This was a small pilot study and consent was not obtained to share data.